CLINICAL TRIAL: NCT04189601
Title: Complement Activation in the Lysosomal Storage Disorders
Acronym: CATALYST
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator Dr. Thomas Barbour passed away.
Sponsor: Melbourne Health (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: Royal_Melbourne
Record Dates: First submitted 2019-12-01; First posted 2019-12-06 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease; Gaucher Disease; Niemann-Pick Disease, Type C; Lysosomal Storage Diseases
Keywords: complement
MeSH Terms: conditions — Fabry Disease; Gaucher Disease; Niemann-Pick Disease, Type C; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study subjects: Patients with Fabry disease, Gaucher disease, or Niemann-Pick disease, type D
  Interventions: Diagnostic Test: Complement measurements
- Controls: Age- and sex-matched to Study subjects
  Interventions: Diagnostic Test: Complement measurements

INTERVENTIONS:
Diagnostic Test: Complement measurements — Blood and urine tests to assess the complement activation state

SUMMARY:
The lysosomal storage disorders (LSDs) are monogenic disorders associated with inflammation affecting multiple organs, and early death. Few treatments are available that can modify the disease course, and there is an urgent need to identify new steps in pathogenesis that can be targeted therapeutically. The complement system is novel and highly plausible as a primary driver of inflammation and cellular injury in the LSDs. This study assesses the complement activation state in patients with Fabry disease (FD), Gaucher disease (GD) and Niemann-Pick disease, type C (NPC), with comparison to healthy controls. This has the potential for immense clinical benefit through targeted complement inhibition across the full spectrum of lysosomal storage disorders, in which key pathophysiological processes including the inflammatory response to lysosomally 'stored' materials are shared.

DETAILED DESCRIPTION:
This is a single-centre, cross-sectional observational study in patients >16 years of age diagnosed with FD, GD or NPC. The research hypotheses of this study are:

1. That complement is excessively activated, including at the specifically complement C5 level, in patients with the lysosomal storage disorders FD, GD and NPC.
2. That complement activation drives tissue injury in the LSDs via downstream effector mechanisms including membrane attach complex (MAC/C5b-9)-mediated cytotoxicity and C5aR-mediated inflammation.

The study aims to show enhanced complement activation, including at the C5 level, in patients with FD, GD and NPC compared to healthy controls.

The research assays for this study include the primary outcome measure of plasma soluble C5b-9 (sC6b-9) levels measured using ELISA. This assay measures the degree to which ongoing C5 activation Is occurring in vivo based on sensitive detection in plasma of the key activation product C5b-9. The assay would be expected to show elevated plasma sC5b-9 levels in patients with the glycosphingolipidoses compared to disease-free controls, as was previously demonstrated in patient cohorts of atypical haemolytic uraemia syndrome (aHUS) and C3 glomerulopathy (C3G). Additional complement activation products will be assessed as secondary endpoints including plasma C3a and C5a levels by ELISA, and intracellular leukocyte C5a concentration as a marker of systemic C5a generation and C5aR1 expression.

ELIGIBILITY:
Inclusion Criteria:

* All consenting patients with a prior diagnosis of FD, GD or NPC will be included in the study. Control participants will be healthy volunteers.

Exclusion Criteria:

* Patients who are unable to provide consent or to perform a blood or urine test will be excluded.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consenting patients with FD, GD or NPC, and age and sex-matched controls
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-02-26 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in soluble C5b-9 | At baseline
  Difference in sC5b-9 between Subjects and Controls at a single timepoint up to 8 months

SECONDARY OUTCOMES:
Other complement biomarkers | Difference in C3a and C5a between Subjects and Controls at a single timepoint up to 8 months
  Serum C3a and C5a

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Barbour, MBBS, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD sharing